CLINICAL TRIAL: NCT04446585
Title: A Cluster Randomized Clinical Trial of Strategic AED Deployment in High-risk Residential Areas Combined With Activation of Local Residents
Brief Title: Cardiac Arrest in Residential Areas With Mobile First-responder Activation
Acronym: CARAMBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: TrygFonden, Denmark (Industry); Zoll Medical Corporation (Industry); Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Fredrik Folke, M.D., PhD, Professor, Emergency Medical Services, Capital Region, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Suddan cardiac arrest; Heart Arrest; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest; Heart Diseases; Cardiovascular Diseases | interventions — Defibrillators; Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, treatment allocation is not masked to rescuers or patients. The steering committee will, during the study, receive information on total numbers of arrests and overall success of providing defibrillation. The steering committee will not receive information on whether defibrillation took place in areas allocated to intervention or no intervention. Only the safety committee will have access to all information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control sites (No Intervention): * For all 1-1-2 calls with suspected cardiac arrest to the emergency dispatch center will activate a two-tiered response consisting of dispatch of an ambulance with an emergency medical technician, a physician-staffed mobile emergency care unit, and citizen first responders through the Heart Runner app.
  * The medical dispatcher offers telephone assisted cardiopulmonary resuscitation (CPR) to bystanders. Furthermore, if more than two bystanders are present and an AED is accessible within 1½ minute travel distance (depending on the type of terrain), then one bystander is guided to localize and retrieve the AED.
- Intervention sites (Experimental): As a supplement to the standard care as described in the control arm, the following will be supplied:
  * Strategical deployment of AEDs with 24:7 availability and 1½ minute walking distance to every residence within the area. The AEDs will be registered with the AED network and thus linked to the emergency dispatch center.
  * The emergency dispatch center will retrieve data from used AEDs.
  * For each interventional area, approximately 120 residents will receive a course in CPR and AED use and subsequently be recruited as citizen responders so that they can be activated through the HeartRunner app in case of a nearby cardiac arrest.
  Interventions: Device: Automated External Defibrillator (AED); Other: Training in cardiopulmonary resuscitation and AED use; Other: Activation of citizen responders

INTERVENTIONS:
Device: Automated External Defibrillator (AED) — Deployment of AEDs
  Arms: Intervention sites
Other: Training in cardiopulmonary resuscitation and AED use — Residents will undergo 30-minute courses at study start and if needed during the trial period. During the course they will also be recruited as citizen responders
  Arms: Intervention sites
Other: Activation of citizen responders — Citizen responders will be activated in case of suspected cardiac arrest through the heart runner app.
  Arms: Intervention sites

SUMMARY:
The study aims to increase proportions of bystander defibrillation during out-of-hospital cardiac arrest (hereof referred to as cardiac arrest) in residential areas with a high density of cardiac arrests. The intervention consists of Automated External Defibrillators (AEDs) and residents' involvement in resuscitation through training and enrollment as citizen responders.

DETAILED DESCRIPTION:
Survival decreases by 10% for every minute that passes after a cardiac arrest until defibrillation. Despite an increasing number of available AEDs, survival and defibrillation rates in residential areas remain poor. Efforts to increase bystander defibrillation has the potential to improve survival. Through the strategic deployment of AEDs, training, and recruitment of residents as citizen responders, we aim to improve proportions of bystander defibrillation and 30-day survival in densely populated residential areas with a high density of cardiac arrests.

ELIGIBILITY:
Inclusion Criteria:

* All witnessed cardiac arrests recognized registered in the Danish Cardiac Arrest Registry occurring within the study sites. This excludes non witnessed cardiac arrests.
* Witnessed cardiac arrest
* Non-traumatic etiology, this excludes intoxication, drowning or suicide.

Exclusion Criteria:

* Cardiac arrest occurring in a nursing home
* Cardiac arrest not treated by the EMS due to ethical reasons or obvious signs of death
* Not true cardiac arrest (suspected, but not verified)
* Cardiac arrests witnessed by the emergency medical personnel

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Bystander defibrillation | Up to five years after implementation of the intervention
  Proportion of bystander defibrillation of witnessed cardiac arrests

SECONDARY OUTCOMES:
30-day survival | 30 days after date of cardiac arrest
  Proportion of patients alive 30 days after date of cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Folke, MD, PhD, Principal Investigator — EMS Copenhagen; Carolina M Hansen, MD, PhD, Principal Investigator — EMS Copenhagen
Locations (1):
- Emergency Medical Services Copenhagen, Ballerup Municipality, The Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juul Grabmayr A, Malta Hansen C, Bo N, Sheikh AP, Hassager C, Ersboll A, Kjaergaard J, Lippert F, Tjornhoj-Thomsen T, Gislason G, Torp-Pedersen C, Folke F. Community intervention to improve defibrillation before ambulance arrival in residential neighbourhoods with a high risk of out-of-hospital cardiac arrest: study protocol of a cluster-randomised trial (the CARAMBA trial). BMJ Open. 2023 Oct 10;13(10):e073541. doi: 10.1136/bmjopen-2023-073541. PMID 37816557

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04446585/Prot_SAP_001.pdf